CLINICAL TRIAL: NCT05785195
Title: Study on the Mechanism of Inhaled Nitric Oxide in the Treatment of Patients With Chronic Obstructive Pulmonary Disease (COPD) Complicated With Pulmonary Hypertension
Brief Title: A Mechanistic Study of Inhaled Nitric Oxide in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ting YANG (Other)
Collaborators: Novlead Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ting YANG, Clinical Professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-HX-110
Record Dates: First submitted 2023-02-17; First posted 2023-03-27 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled Nitric Oxide (iNO) (Experimental): iNO 20ppm，≥8 hours/day for 3 days
  Interventions: Device: Nitric Oxide Generation and Delivery System

INTERVENTIONS:
Device: Nitric Oxide Generation and Delivery System — The Nitric Oxide Generation and Delivery System is used to deliver nitric oxide for inhalation therapy into the inspiratory limb of the patient breathing circuit in a way that provides a constant concentration of nitric oxide (NO), as set by the user, to the patient throughout the inspired breath.

SUMMARY:
There is a lack of effective treatments for chronic obstructive pulmonary disease (COPD) complicated with pulmonary hypertension. Previous studies have found that inhaled nitric oxide (iNO) can reduce pulmonary artery pressure and improve exercise capacity in COPD with pulmonary hypertension patients. However, the specific mechanism is unclear. The study aims to evaluate pulmonary ventilation/perfusion, pulmonary artery pressure, oxygenation, symptoms and quality of life in COPD with pulmonary hypertension patients after short-term treatment with iNO. Observing a series of pathophysiological changes caused by the treatment of pulmonary hypertension with iNO in COPD, the investigators hope to provide new theoretical basis and research ideas.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years, ≤ 75 years
2. Currently smoking or former smokers with at least 10 pack-years of tobacco cigarette smoking history
3. Diagnosis of moderate and severe COPD by the Global initiative for chronic Obstructive Lung Disease (GOLD) 2022 criteria: A post-bronchodilatory forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 0.7, and 30%< FEV1 < 80% predicted
4. Echocardiogram with technical adequacy demonstrating with Pulmonary Hypertension: Tricuspid regurgitation velocity (TRV) > 2.8 m/s or pulmonary arterial systolic pressure (sPAP) ≥38mmHg
5. Signed informed consent prior to the initiation of any study mandated procedures or assessments

Exclusion Criteria:

1. Experienced an exacerbation requiring start of or increase in systemic oral corticosteroid therapy during the last month
2. Treatment with antibiotics
3. Respiratory failure requiring supplemental oxygen therapy
4. A diagnosis of Interstitial lung disease, asthma, tuberculosis, bronchiectasis, pneumonia, lung cancer, pulmonary embolism, or other non-COPD respiratory disease
5. Any history of lung resection
6. Left ventricular dysfunction: left ventricular ejection fraction (LVEF) < 40%
7. Clinically significant valvular heart disease, including aortic valvular disease (moderate or greater aortic stenosis or regurgitation) and/or mitral valve disease (moderate or greater mitral stenosis or regurgitation), or status post mitral valve replacement
8. Use within 30 days of screening or current use of approved PH medications such as sildenafil, bosentan or prostacyclines
9. Neuromuscular disease or musculoskeletal injuries that unable to complete exercise trials
10. Use of investigational drugs or devices within 30 days prior to enrollment into the study
11. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Ventilation-perfusion ratio | Baseline, Minutes 30
  Change in ventilation-perfusion ratio (V/Q) from Baseline after treatment with iNO, measured by pulmonary ventilation/perfusion imaging
Tricuspid regurgitation velocity (TRV) | Baseline, Day 3
  Change in TRV from Baseline after treatment with iNO, measured by echocardiogram
Pulmonary arterial systolic pressure (sPAP) | Baseline, Day 3
  Change in sPAP from Baseline after treatment with iNO, measured by echocardiogram

SECONDARY OUTCOMES:
Percutaneous arterial oxygen saturation (SpO2) | Baseline, Day 3
  Change in SpO2 from Baseline after treatment with iNO
Pulmonary function:Forced expiratory volume in 1 second（FEV1） | Baseline, Day 3
  Change in FEV1 from Baseline after treatment with iNO
Pulmonary function: Forced vital capacity （FVC） | Baseline, Day 3
  Change in FVC from Baseline after treatment with iNO
Pulmonary function: FEV1/FVC | Baseline, Day 3
  Change in ratio of FEV1 and FVC (FEV1/FVC) from Baseline after treatment with iNO
Pulmonary function: Diffusion lung capacity for carbon monoxide（DLCO) | Baseline, Day 3
  Change in DLCO from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Maximal oxygen uptake（VO2max） | Baseline, Day 3
  Change in VO2max from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Anaerobic threshold（AT） | Baseline, Day 3
  Change in AT from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Minute ventilation-to-carbon dioxide output（VE/VCO2） | Baseline, Day 3
  Change in VE/VCO2 from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Physiological dead space ventilation (physiological deadspace volume/tidal volume, Vd/Vt) | Baseline, Day 3
  Change in Vd/Vt from Baseline after treatment with iNO
Six-minute walk distance (6MWD) | Baseline, Day 3
  Change in 6MWD from Baseline after treatment with iNO
Arterial blood gas: Arterial partial pressure of oxygen (PaO2) | Baseline, Day 3
  Change in PaO2 from Baseline after treatment with iNO
Arterial blood gas: Arterial partial pressure of carbon dioxide (PaCO2) | Baseline, Day 3
  Change in PaCO2 from Baseline after treatment with iNO
Arterial blood gas: Alveolar-arterial oxygen partial pressure difference (A-aDO2) | Baseline, Day 3
  Change in A-aDO2 from Baseline after treatment with iNO
Life quality and symtom severity questionnaires: COPD assessment test (CAT) | Baseline, Day 3
  Change in CAT scores (0-40 scores, higher scores mean a worse outcome) from Baseline after treatment with iNO
Life quality and symtom severity questionnaires: Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline, Day 3
  Change in (mMRC) Dyspnea Scale scores (0-4 scores, higher scores mean a worse outcome) from Baseline after treatment with iNO
Life quality and symtom severity questionnaires: Saint George Respiratory Questionnaire (SGRQ) | Baseline, Day 3
  Change in SGRQ scores (0-100 scores, higher scores mean a worse outcome) from Baseline after treatment with iNO
Adverse events | Baseline up to Day 3
  Incidence of adverse events = Number of subjects with adverse events/Total number of subjects in treatment×100%

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No